CLINICAL TRIAL: NCT01001299
Title: A Multi-center, Open-label, Study to Investigate the Pharmacokinetic Interaction of RO5185426 With a "Cocktail" of Five Probe Drugs for CYP450 Dependent Metabolism in Patients With Previously Treated and Untreated Metastatic Melanoma
Brief Title: A Pharmacokinetic Study of RO5185426 in Combination With a Drug Cocktail in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP22676
Record Dates: First submitted 2009-10-21; First posted 2009-10-26 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-06

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Drug cocktail; Drug: RO5185426

INTERVENTIONS:
Drug: Drug cocktail — Drug cocktail (caffeine, warfarin + vitamin K, omeprazole, dextromethorphan, midazolam) orally once daily, day 1 and day 20
Drug: RO5185426 — 960 mg orally twice daily

SUMMARY:
This open-label single-arm study will evaluate the effect of RO5185426 [RG7204; PLEXXIKON: PLX4032] on the pharmacokinetics of five CYP450 substrates (caffeine, warfarin + vitamin K, omeprazole, dextromethorphan, midazolam) administered as a drug cocktail to patients with metastatic melanoma. The study will also evaluate efficacy and safety of RO5185426. On day 1, patients will receive the drug cocktail. On days 6 to 19, patients will receive RO5185426 twice daily. On day 20, patients will receive RO5185426 and the drug cocktail and on days 21 to 25, patients will receive RO5185426. Assessments will be made at regular intervals during the dosing periods and at follow-up. Patients may continue on study treatment (RO5185426) until the development of progressive disease or unacceptable toxicity. Target sample size <50.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient >/= 18 years of age
* Malignant melanoma (Stage IV, AJCC)
* Patients who are treatment-naive or have received prior systemic treatments for metastatic melanoma. Time elapsed between previous treatment for metastatic disease and first administration of study drug must be at least 28 days
* Positive tested for BRAF mutation
* Patients must not be poor metabolizers of CYP450 enzymes 2C9, 2C19, or 2D6 as determined by genotyping
* Measurable disease by RECIST criteria
* Negative pregnancy test; for fertile men and women, effective contraception during treatment and for 6 months after completion

Exclusion Criteria:

* Active CNS lesions on CT/MRI within 28 days prior to enrollment
* History of known spinal cord compression, or carcinomatous meningitis
* Severe cardiovascular disease within 6 months prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - UCLA - School of Medicine, Los Angeles, California
  - Massachusetts General Hospital;Hematology/ Oncology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas

REFERENCES:
- [Derived] Su F, Viros A, Milagre C, Trunzer K, Bollag G, Spleiss O, Reis-Filho JS, Kong X, Koya RC, Flaherty KT, Chapman PB, Kim MJ, Hayward R, Martin M, Yang H, Wang Q, Hilton H, Hang JS, Noe J, Lambros M, Geyer F, Dhomen N, Niculescu-Duvaz I, Zambon A, Niculescu-Duvaz D, Preece N, Robert L, Otte NJ, Mok S, Kee D, Ma Y, Zhang C, Habets G, Burton EA, Wong B, Nguyen H, Kockx M, Andries L, Lestini B, Nolop KB, Lee RJ, Joe AK, Troy JL, Gonzalez R, Hutson TE, Puzanov I, Chmielowski B, Springer CJ, McArthur GA, Sosman JA, Lo RS, Ribas A, Marais R. RAS mutations in cutaneous squamous-cell carcinomas in patients treated with BRAF inhibitors. N Engl J Med. 2012 Jan 19;366(3):207-15. doi: 10.1056/NEJMoa1105358. PMID 22256804

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The five probe parent drugs used in the study were caffeine (metabolite: paraxanthine), S-warfarin (no metabolite), omeprazole (metabolite: hydroxy [OH]-omeprazole), dextromethorphan (metabolite: dextrorphan), and midazolam (metabolite: OH-midazolam).
Groups:
- Vemurafenib: Single oral doses of 5 probe drugs (caffeine 200 milligrams [mg] tablet, warfarin 10 mg tablet [with Vitamin K 10 mg {2*5 mg tablets}], omeprazole 40 mg capsule, dextromethorphan 30 mg syrup, and midazolam 0.075 milligrams per kilogram [mg/kg] syrup) on Day 1, followed by 5-day washout. Vemurafenib (RO5185426) 960 mg (4*240 mg film-coated tablets) orally twice daily on Day 6 to Day 19. Single oral doses of 5 probe drugs co-administered with vemurafenib 960 mg on Day 20, followed by vemurafenib 960 mg orally twice daily up to Day 28 and then vemurafenib 960 mg orally twice daily continuously in 28-day cycles until disease progression, toxicity, withdrawal of consent, loss to follow-up, or death (whichever occurred first).
Period: Overall Study
Arm/Group | Vemurafenib
Started | 25
Completed | 0
Not Completed | 25
Not completed — Insufficient Therapeutic Response | 20
Not completed — Adverse event or Intercurrent Illness | 1
Not completed — Death | 1
Not completed — Began Taking Commercially Available Drug | 2
Not completed — Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants.
Groups:
- Vemurafenib: Single oral doses of 5 probe drugs (caffeine 200 mg tablet, warfarin 10 mg tablet [with Vitamin K 10 mg {2*5 mg tablets}], omeprazole 40 mg capsule, dextromethorphan 30 mg syrup, and midazolam 0.075 mg/kg syrup) on Day 1, followed by 5-day washout. Vemurafenib 960 mg (4*240 mg film-coated tablets) orally twice daily on Day 6 to Day 19. Single oral doses of 5 probe drugs co-administered with vemurafenib 960 mg on Day 20, followed by vemurafenib 960 mg orally twice daily up to Day 28 and then vemurafenib 960 mg orally twice daily continuously in 28-day cycles until disease progression, toxicity, withdrawal of consent, loss to follow-up, or death (whichever occurred first).
Arm/Group | Vemurafenib
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratio of Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Observed Sampling Time (AUC[0-last]) of Probe Parent Drugs
Description: AUC(0-last) was defined as the area under the plasma concentration-time curve calculated using the linear trapezoidal rule from time zero to the last observed sampling time. To assess the potential for drug-drug interactions, the geometric mean ratios and corresponding 90 percent (%) confidence interval (CI) of AUC(0-last) of parent probe drug before (Day 1) and after treatment with vemurafenib (Day 20) was calculated. Ratio and corresponding 90% CI of AUC(0-last) (Day 20/Day 1) for each of the 5 probe drugs is reported.
Time Frame: Day 1, 20: 0, 1, 3, 4, 6, 8, 24 hours, additionally for caffeine 0.5, 1.5, 2, 12, 18, 48, 72, 96, 120,dextromethorphan 0.5, 1.5, 2, 12, 18, 48,midazolam 0.08, 0.25, 0.5, 0.75, 2, 10,omeprazole 0.5, 1.5, 2, 2.5, 12, 18,S-warfarin 12, 48, 72, 96, 120 hours
Population: Primary pharmacokinetic (PK) population: all participants who received all planned doses of vemurafenib without dose modification/interruption up to Day 25 and all doses of 5 cocktail probes, without major protocol violation. Number of Participants Analyzed=participants evaluable for this outcome; n=participants evaluable for specified category.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
ratio
  Caffeine (n = 19) | 2.56 [2.24 to 2.93]
  Dextromethorphan (n = 20) | 1.47 [1.21 to 1.78]
  Midazolam (n = 20) | 0.61 [0.50 to 0.74]
  Omeprazole (n = 20) | 1.13 [0.92 to 1.37]
  S-warfarin (n = 20) | 1.18 [1.12 to 1.24]

2. Primary Outcome: Geometric Mean Ratio of Maximum Plasma Concentration (Cmax) of Probe Parent Drugs
Description: To assess the potential for drug-drug interactions, the geometric mean ratios and corresponding 90% CI of Cmax of parent probe drug before (Day 1) and after treatment with vemurafenib (Day 20) was calculated. Ratio and corresponding 90% CI of Cmax (Day 20/Day 1) for each of the 5 probe drugs is reported.
Time Frame: as for outcome 1
Population: Primary PK analysis population. Number of Participants Analyzed = participants evaluable for this outcome and n = participants evaluable for specified category.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
ratio
  Caffeine (n = 19) | 1.05 [0.98 to 1.13]
  Dextromethorphan (n = 20) | 1.36 [1.07 to 1.72]
  Midazolam (n = 20) | 0.65 [0.54 to 0.78]
  Omeprazole (n = 20) | 1.17 [0.92 to 1.49]
  S-warfarin (n = 20) | 1.00 [0.93 to 1.08]

3. Primary Outcome: Geometric Mean Ratio of AUC(0-last) and Cmax of Metabolites of Probe Parent Drugs
Description: AUC(0-last) was defined as the area under the plasma concentration-time curve calculated using the linear trapezoidal rule from time zero to the last observed sampling time. To assess the potential for drug-drug interactions, the geometric mean ratios and corresponding 90% CI of AUC(0-last) and Cmax of metabolites of parent probe drug before (Day 1) and after treatment with vemurafenib (Day 20) was calculated. Ratio and corresponding 90% CI of AUC(0-last) and Cmax (Day 20/Day 1) for each of the 4 probe drug metabolites is reported (paraxanthine [caffeine metabolite], dextrorphan [dextromethorphan metabolite], OH-midazolam [midazolam metabolite], OH-omeprazole (omeprazole metabolite); S-warfarin does not have a metabolite).
Time Frame: Day 1, 20: 0, 1, 3, 4, 6, 8, 24 hours, additionally for paraxanthine 0.5, 1.5, 2, 12, 18, 48, 72, 96, 120, dextrorphan 0.5, 1.5, 2, 12, 18, 48, OH-midazolam 0.08, 0.25, 0.5, 0.75, 2, 10, OH-omeprazole 0.5, 1.5, 2, 2.5, 12, 18 hours
Population: as for outcome 2
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
ratio
  Paraxanthine - AUC(0-last) (n = 19) | 1.15 [0.98 to 1.36]
  Paraxanthine - Cmax (n = 19) | 0.60 [0.53 to 0.68]
  Dextrorphan - AUC(0-last) (n = 20) | 1.46 [1.22 to 1.75]
  Dextrorphan - Cmax (n = 20) | 1.21 [0.97 to 1.51]
  OH-Midazolam - AUC(0-last) (n = 20) | 1.34 [1.17 to 1.54]
  OH-Midazolam - Cmax (n = 20) | 1.23 [1.04 to 1.44]
  OH-Omeprazole - AUC(0-last) (n = 20) | 1.16 [1.06 to 1.28]
  OH-Omeprazole - Cmax (n = 20) | 1.01 [0.87 to 1.18]

4. Primary Outcome: AUC(0-last) and Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC[0-inf]) of Probe Parent Drugs and Their Metabolites on Day 1
Description: AUC(0-last) was defined as the area under the plasma concentration-time curve calculated using the linear trapezoidal rule from time zero to the last observed sampling time. AUC(0-inf) was defined as the area under the plasma concentration-time curve calculated using the linear trapezoidal rule from time zero extrapolated to infinity. Timeframe reported for parent probe drug is also applicable for their metabolite except S-warfarin, as S-warfarin does not have a metabolite.
Time Frame: Day 1: 0, 1, 3, 4, 6, 8, 24 hours, additionally for caffeine 0.5, 1.5, 2, 12, 18, 48, 72, 96, 120,dextromethorphan 0.5, 1.5, 2, 12, 18, 48,midazolam 0.08, 0.25, 0.5, 0.75, 2, 10,omeprazole 0.5, 1.5, 2, 2.5, 12, 18,S-warfarin 12, 48, 72, 96, 120 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
nanograms*hour per milliliter (ng*hr/mL)
  Caffeine - AUC(0-last) (n = 19) | 56350.1 (24744.07)
  Caffeine - AUC(0-inf) (n = 19) | 58337.5 (25287.72)
  Paraxanthine - AUC(0-last) (n = 19) | 45584.3 (15667.21)
  Paraxanthine - AUC(0-inf) (n = 19) | 47589.5 (16667.35)
  S-Warfarin - AUC(0-last) (n = 20) | 14964.5 (4566.80)
  S-Warfarin - AUC(0-inf) (n = 20) | 17832.5 (6785.62)
  Omeprazole - AUC(0-last) (n = 20) | 3110.4 (2956.30)
  Omeprazole - AUC(0-inf) (n = 20) | 3181.0 (3107.71)
  OH-Omeprazole - AUC(0-last) (n = 20) | 1187.0 (353.49)
  OH-Omeprazole - AUC(0-inf) (n = 20) | 1215.3 (398.67)
  Dextromethorphan - AUC(0-last) (n = 20) | 28.37 (45.677)
  Dextromethorphan - AUC(0-inf) (n = 20) | 29.79 (48.159)
  Dextrorphan - AUC(0-last) (n = 20) | 26.76 (19.368)
  Dextrorphan - AUC(0-inf) (n = 20) | 29.34 (19.865)
  Midazolam - AUC(0-last) (n = 20) | 100.18 (53.949)
  Midazolam - AUC(0-inf) (n = 20) | 103.57 (55.767)
  OH-Midazolam - AUC(0-last) (n = 20) | 42.96 (22.197)
  OH-Midazolam - AUC(0-inf) (n = 20) | 44.70 (22.632)

5. Primary Outcome: AUC(0-last) and AUC(0-inf) of Probe Parent Drugs and Their Metabolites on Day 20
Description: as for outcome 4
Time Frame: Day 20: 0, 1, 3, 4, 6, 8, 24 hours, additionally for caffeine 0.5, 1.5, 2, 12, 18, 48, 72, 96, 120,dextromethorphan 0.5, 1.5, 2, 12, 18, 48,midazolam 0.08, 0.25, 0.5, 0.75, 2, 10,omeprazole 0.5, 1.5, 2, 2.5, 12, 18,S-warfarin 12, 48, 72, 96, 120 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
ng*hr/mL
  Caffeine - AUC(0-last) (n = 19) | 140991.9 (56983.62)
  Caffeine - AUC(0-inf) (n = 19) | 161490.6 (81139.12)
  Paraxanthine - AUC(0-last) (n = 19) | 51344.3 (14888.54)
  Paraxanthine - AUC(0-inf) (n = 19) | 55060.5 (15481.99)
  S-Warfarin - AUC(0-last) (n = 20) | 17804.4 (5956.35)
  S-Warfarin - AUC(0-inf) (n = 20) | 22233.3 (9485.43)
  Omeprazole - AUC(0-last) (n = 20) | 3155.6 (3090.03)
  Omeprazole - AUC(0-inf) (n = 20) | 3224.9 (3200.67)
  OH-Omeprazole - AUC(0-last) (n = 20) | 1370.2 (370.57)
  OH-Omeprazole - AUC(0-inf) (n = 20) | 1409.9 (398.39)
  Dextromethorphan - AUC(0-last) (n = 20) | 39.33 (56.972)
  Dextromethorphan - AUC(0-inf) (n = 20) | 41.56 (62.027)
  Dextrorphan - AUC(0-last) (n = 20) | 37.74 (23.402)
  Dextrorphan - AUC(0-inf) (n = 20) | 40.85 (24.333)
  Midazolam - AUC(0-last) (n = 20) | 67.70 (50.773)
  Midazolam - AUC(0-inf) (n = 20) | 69.82 (52.705)
  OH-Midazolam - AUC(0-last) (n = 20) | 59.78 (34.419)
  OH-Midazolam - AUC(0-inf) (n = 20) | 64.25 (35.604)

6. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 8, 12, and 24 Hours (AUC[0-8], AUC[0-12], AUC[0-24]) of Vemurafenib
Description: Area under the plasma concentration-time curve calculated using the linear trapezoidal rule from time zero to 8, 12, and 24 hours (AUC[0-8], AUC[0-12], AUC[0-24], respectively).
Time Frame: 0, 0.5, 1, 2, 4, 8, 12, 13, 14, 16, 18, 24 hours on Day 19
Population: Primary PK analysis population.
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter (mcg*h/mL)
Arm/Group | Vemurafenib
Number analyzed (Participants) | 21
micrograms*hour/milliliter (mcg*h/mL)
  AUC(0-8) | 422 (121)
  AUC(0-12) | 601 (170)
  AUC(0-24) | 1176 (368)

7. Primary Outcome: Cmax of Probe Parent Drugs and Their Metabolites on Day 1
Description: Timeframe reported for parent probe drug is also applicable for their metabolite except S-warfarin as S-warfarin does not have a metabolite.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
nanograms per milliliter (ng/mL)
  Caffeine - Cmax (n = 19) | 4768.9 (1108.43)
  Paraxanthine - Cmax (n = 19) | 1839.1 (477.75)
  S-Warfarin - Cmax (n = 20) | 469.4 (127.22)
  Omeprazole - Cmax (n = 20) | 913.7 (610.63)
  OH-Omeprazole - Cmax (n = 20) | 331.3 (127.60)
  Dextromethorphan - Cmax (n = 20) | 3.38 (4.236)
  Dextrorphan - Cmax (n = 20) | 6.49 (5.041)
  Midazolam - Cmax (n = 20) | 41.88 (29.197)
  OH-Midazolam - Cmax (n = 20) | 18.54 (9.938)

8. Primary Outcome: Cmax of Probe Parent Drugs and Their Metabolites on Day 20
Description: as for outcome 7
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
ng/mL
  Caffeine - Cmax (n = 19) | 4990.5 (1005.33)
  Paraxanthine - Cmax (n = 19) | 1154.9 (446.30)
  S-Warfarin - Cmax (n = 20) | 468.3 (115.63)
  Omeprazole - Cmax (n = 20) | 945.8 (535.41)
  OH-Omeprazole - Cmax (n = 20) | 348.7 (168.43)
  Dextromethorphan - Cmax (n = 20) | 4.19 (5.342)
  Dextrorphan - Cmax (n = 20) | 7.10 (4.332)
  Midazolam - Cmax (n = 20) | 26.18 (13.811)
  OH-Midazolam - Cmax (n = 20) | 22.06 (10.969)

9. Primary Outcome: Cmax of Vemurafenib
Time Frame: 0, 0.5, 1, 2, 4, 8, 12, 13, 14, 16, 18, 24 hours on Day 19
Population: Primary PK analysis population.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Vemurafenib
Number analyzed (Participants) | 21
micrograms per milliliter (mcg/mL) | 61.7 (17.2)

10. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Probe Parent Drugs and Their Metabolites on Day 1
Description: as for outcome 7
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
hours
  Caffeine - Tmax (n = 19) | 1.00 [1.00 to 3.00]
  Paraxanthine - Tmax (n = 19) | 8.00 [4.00 to 24.00]
  S-Warfarin - Tmax (n = 20) | 3.00 [1.00 to 6.00]
  Omeprazole - Tmax (n = 20) | 3.00 [1.00 to 8.00]
  OH-Omeprazole - Tmax (n = 20) | 3.00 [1.00 to 8.00]
  Dextromethorphan - Tmax (n = 20) | 1.50 [0.50 to 3.00]
  Dextrorphan - Tmax (n = 20) | 1.50 [0.50 to 4.00]
  Midazolam - Tmax (n = 20) | 0.50 [0.25 to 2.00]
  OH-Midazolam - Tmax (n = 20) | 0.50 [0.25 to 2.00]

11. Primary Outcome: Tmax of Probe Parent Drugs and Their Metabolites on Day 20
Description: as for outcome 7
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
hours
  Caffeine - Tmax (n = 19) | 2.00 [1.00 to 122.00]
  Paraxanthine - Tmax (n = 19) | 24.00 [8.00 to 122.00]
  S-Warfarin - Tmax (n = 20) | 3.00 [1.00 to 8.00]
  Omeprazole - Tmax (n = 20) | 2.5 [1.0 to 8.0]
  OH-Omeprazole - Tmax (n = 20) | 3.00 [1.00 to 8.00]
  Dextromethorphan - Tmax (n = 20) | 1.50 [0.50 to 3.00]
  Dextrorphan - Tmax (n = 20) | 1.50 [1.00 to 3.00]
  Midazolam - Tmax (n = 20) | 0.50 [0.25 to 1.05]
  OH-Midazolam - Tmax (n = 20) | 0.50 [0.25 to 2.25]

12. Primary Outcome: Tmax of Vemurafenib
Time Frame: 0, 0.5, 1, 2, 4, 8, 12, 13, 14, 16, 18, 24 hours on Day 19
Population: Primary PK analysis population.
Measure: Median (Full Range); unit: hours
Arm/Group | Vemurafenib
Number analyzed (Participants) | 21
hours | 3.10 [0.00 to 26.1]

13. Primary Outcome: Trough Plasma Concentration (Cmin) of Vemurafenib
Time Frame: Before morning dose (0 hour) on Day 19
Population: Primary PK analysis population. Here, number of participants analyzed signifies participants with evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
mcg/mL | 54.5 (18.55)

14. Primary Outcome: Apparent Elimination Half-Life in Plasma (t1/2) of Probe Parent Drugs and Their Metabolites on Day 1
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Primary PK analysis population. Number of Participants Analyzed = participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
hours
  Caffeine - t1/2 | 6.7 (3.42)
  Paraxanthine - t1/2 | 18.5 (24.84)
  S-Warfarin - t1/2 | 42.3 (18.16)
  Omeprazole - t1/2 | 2.0 (1.65)
  OH-Omeprazole - t1/2 | 2.6 (1.90)
  Dextromethorphan - t1/2 | 9.08 (2.211)
  Dextrorphan - t1/2 | 4.08 (1.612)
  Midazolam - t1/2 | 5.06 (1.787)
  OH-Midazolam - t1/2 | 5.46 (2.749)

15. Primary Outcome: t1/2 of Probe Parent Drugs and Their Metabolites on Day 20
Description: as for outcome 7
Time Frame: as for outcome 5
Population: Primary PK analysis population. Number of Participants Analyzed = participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
hours
  Caffeine - t1/2 | 20.6 (11.94)
  Paraxanthine - t1/2 | 35.3 (16.57)
  S-Warfarin - t1/2 | 47.4 (21.30)
  Omeprazole - t1/2 | 2.6 (2.27)
  OH-Omeprazole - t1/2 | 3.2 (2.09)
  Dextromethorphan - t1/2 | 8.24 (2.884)
  Dextrorphan - t1/2 | 4.42 (1.625)
  Midazolam - t1/2 | 4.00 (1.648)
  OH-Midazolam - t1/2 | 7.94 (4.581)

16. Primary Outcome: Apparent Plasma Clearance (CL/F) of Probe Parent Drugs on Day 1
Description: Drug clearance was a quantitative measure of the rate at which a drug substance was removed from the body. Clearance obtained after oral dose was influenced by the fraction of the dose absorbed.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliters per hour (mL/h)
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
milliliters per hour (mL/h)
  Caffeine - CL/F (n = 19) | 4.2 (2.03)
  S-Warfarin - CL/F (n = 20) | 622.4 (184.13)
  Omeprazole - CL/F (n = 20) | 0.035 (0.035)
  Dextromethorphan - CL/F (n = 20) | 4108.04 (4117.517)
  Midazolam - CL/F (n = 20) | 72199.55 (35742.230)

17. Primary Outcome: CL/F of Probe Parent Drugs on Day 20
Description: as for outcome 16
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Vemurafenib
Number analyzed (Participants) | 20
mL/h
  Caffeine - CL/F (n = 19) | 1.6 (0.77)
  S-Warfarin - CL/F (n = 20) | 513.5 (168.97)
  Omeprazole - CL/F (n = 20) | 0.027 (0.020)
  Dextromethorphan - CL/F (n = 20) | 2921.59 (3060.460)
  Midazolam - CL/F (n = 20) | 125436.51 (79335.601)

18. Secondary Outcome: Percentage of Participants With a Confirmed Best Overall Response of Complete Response (CR) or Partial Response (PR)
Description: Confirmed best overall response was defined as having best objective response as CR or PR, as assessed by investigator and confirmed at least 28 days after initial response, according to the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1). CR was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must decrease to normal (short axis less than [<] 10 millimeter [mm]). PR was defined as a 30% decrease in the sum of the diameters of the target lesions taking as a reference the baseline sum diameter. Percentage of participants with best overall response of CR or PR are reported.
Time Frame: Screening up to approximately 3.5 years (assessed at Screening, Day 1 of Cycle 3 thereafter Day 1 of every other cycle [every 2 months] and at end of study)
Population: Efficacy population included all enrolled participants who received any vemurafenib and had at least one post-baseline tumor assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 25
percentage of participants | 44

19. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time interval between the date of the earliest qualifying response and the date of disease progression (PD) or death, only for those participants whose best overall response was CR or PR, as assessed by investigator. CR was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must decrease to normal (short axis <10 mm). PR was defined as a 30% decrease in the sum of the diameters of the target lesions taking as a reference the baseline sum diameter. PD was defined as at least 20% increase in the sum of diameters of target lesions compared to Nadir (smallest sum of diameters on-study), unequivocal progression of existing non-target lesions, or presence of new lesion.
Time Frame: as for outcome 18
Population: The data for this outcome measure was not collected as the outcome was removed as per changes in planned analysis (protocol amendment).
Arm/Group | Vemurafenib
Number analyzed (Participants) | 0

20. Secondary Outcome: Time to Response
Description: Time to response was defined as the interval between the date of the first treatment and the date of the first documentation of confirmed CR or PR (as assessed by investigator), whichever occurred first. CR was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must decrease to normal (short axis <10 mm). PR was defined as a 30% decrease in the sum of the diameters of the target lesions taking as a reference the baseline sum diameter.
Time Frame: as for outcome 18
Population: as for outcome 19
Arm/Group | Vemurafenib
Number analyzed (Participants) | 0

21. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined the time interval between the date of the first treatment and the date of progression or death from any cause, whichever occurred first. Deaths that occurred in participants without disease progression were to be considered to be a PFS event on the date of death. Participants who neither progressed nor died were to be censored on the date of the last evaluable tumor assessment prior to the data cutoff date. PD, as assessed by investigator, was defined as at least 20% increase in the sum of diameters of target lesions compared to Nadir (smallest sum of diameters on-study), unequivocal progression of existing non-target lesions, or presence of new lesion.
Time Frame: as for outcome 18
Population: as for outcome 19
Arm/Group | Vemurafenib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last dose of study drug (median treatment duration: 144 days)
Arm/Group | Vemurafenib
Serious Adverse Events (participants affected / at risk) | 12/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=25)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Uveitis (Eye disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cerebrovasular accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=25)
Anaemia (Blood and lymphatic system disorders) | 7
Ear pain (Ear and labyrinth disorders) | 2
Conjunctivitis (Eye disorders) | 2
Dry eye (Eye disorders) | 5
Lacrimation increased (Eye disorders) | 2
Photophobia (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 4
Fatigue (General disorders) | 19
Influenza like illness (General disorders) | 2
Nodule (General disorders) | 2
Oedema peripheral (General disorders) | 7
Pyrexia (General disorders) | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Folliculitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Sunburn (Injury, poisoning and procedural complications) | 4
Blood alkaline phosphatase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 2
Blood creatinine increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 4
Liver function test abnormal (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Weight decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hypovolaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 10
Hyperaesthesia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Gynaecomastia (Reproductive system and breast disorders) | 3
Nipple swelling (Reproductive system and breast disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 4
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 9
Blister (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 12
Dermal cyst (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
The data for 'Duration of Response', 'Time to Response', and 'PFS' was not collected as the outcomes were removed as per changes in planned analysis (protocol amendment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.